CLINICAL TRIAL: NCT03592004
Title: Radiomics of Multiparametric MRI for Neoadjuvant Chemotherapy Outcomes Assessment in Breast Cancer
Brief Title: Radiomics of Mp-MRI Assessing NAC Outcome in Breast Cancer
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Chinese Academy of Sciences (Other Government)
Collaborators: Guangdong Provincial People's Hospital (Other); Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other); Beijing Friendship Hospital (Other); Yunnan Cancer Hospital (Other); Liaoning Cancer Hospital & Institute (Other); First Hospital of China Medical University (Other); Affiliated Hospital of Hebei University (Other)
Responsible Party: Principal Investigator, Zhenyu Liu, Associate Professor, Chinese Academy of Sciences
Other Study IDs: ZLiu
Record Dates: First submitted 2018-06-26; First posted 2018-07-19 (Actual); Last update posted 2018-07-19 (Actual); Status verified 2018-07

CONDITIONS: Breast Cancer; Radiomics; Neoadjuvant Chemotherapy; Multi-parametric MRI
MeSH Terms: conditions — Breast Neoplasms | interventions — Neoadjuvant Therapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (7):
- Guangdong General Hospital
  Interventions: Other: neoadjuvant chemotherapy
- Cancer Hospital Chinese Academy Of Medical Sciences
  Interventions: Other: neoadjuvant chemotherapy
- Beijing Friendship Hospital
  Interventions: Other: neoadjuvant chemotherapy
- Yunnan Cancer Hospital
  Interventions: Other: neoadjuvant chemotherapy
- Liaoning Cancer Hospital
  Interventions: Other: neoadjuvant chemotherapy
- The First Hospital Of China Medical University
  Interventions: Other: neoadjuvant chemotherapy
- Affiliated Hospital Of Hebei University
  Interventions: Other: neoadjuvant chemotherapy

INTERVENTIONS:
Other: neoadjuvant chemotherapy — neoadjuvant chemotherapy

SUMMARY:
This is a single-arm, multicentre study that aims to assess whether Radiomics combining multiparametric MRI and clinical data could be a good predictor of the responses to neoadjuvant chemotherapy in Breast Cancer.

DETAILED DESCRIPTION:
Patients undergo multiparametric MRI (including T2WI, DWI and DCE-MRI) at baseline, after 2 courses of neoadjuvant chemotherapy, and prior to the surgery at least 8 weeks after the treatment procedure. Patients undergo biopsy test in one week after the baseline MRI scan to detect the biomarkers including ER, PR, Her-2 and Ki-67, which can be used to select the treatment plan referring to the NCCN clinical guidelines. After the surgery, responses to neoadjuvant chemotherapy are determined according to the histopathologically examination of the surgically resected specimens.

After completion of treatment procedure, patients are followed up for 5 years.

ELIGIBILITY:
Inclusion Criteria:

* biopsy-proven invasive breast cancer;
* received complete neoadjuvant chemotherapy and no treatment has been done before;
* surgery was performed after completion of neoadjuvant chemotherapy, after which pCR was confirmed by postoperative pathological examination;
* pretreatment MRI data within a month before the start of the treatment was eligible, including T2WI, DWI and DCE-MRI.

Exclusion Criteria:

* not completing neoadjuvant chemoradiotherapy;
* not undergoing surgery at our hospital, or pCR was not assessed;
* lack of T2WI, or DWI or DCE-MRI data;
* insufficient MRI quality to obtain measurements (e.g., owing to motion artifacts);
* had unilateral multifocal cancers, and the correlation between the tumor in MR images and postoperative pathological examination was uncertain.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Chinese
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2018-07-18 (Estimated); Primary Completion 2019-06-01 (Estimated); Study Completion 2022-06-01 (Estimated)

PRIMARY OUTCOMES:
predicting pathological complete response (pCR) or no response (NR) | 20 weeks
  The value of Radiomics of multiparametric MRI in predicting responses to neoadjuvant chemotherapy, including pathological complete response (pCR) and no response (NR).
5 years for Disease free survival | 5 years
  The association between Radiomics of multiparametric MRI and disease free survival (DFS), which defined as the time from the beginning of neoadjuvant chemotherapy to the confirmed time of recurrence or metastatic disease, or death due to any other cause.
5 years for Overall survival | 5 years
  The association between Radiomics of multiparametric MRI and overall survival (OS), which defined as the time from the beginning of neoadjuvant chemotherapy to the death with any causes.

CONTACTS AND LOCATIONS:
Overall Officials: Jie Tian, Doctor, Principal Investigator — Chinese Academy of Sciences
Locations (1):
- Zhenyu Liu, Beijing, China

IPD SHARING:
Plan to Share IPD: No